CLINICAL TRIAL: NCT05931731
Title: Efficacy of Mechanical Interference Versus Neural Mobilization on Ulnar Neuropathy Post Cubital Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: Mechanical Interference Versus Neural Mobilization on Ulnar Neuropathy Post Cubital Tunnel Syndrome
Acronym: CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed tarek Mohamed hefnawy, principle investigator mohamed tarek mohamed hefnawy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003083
Record Dates: First submitted 2023-06-24; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Cubital Tunnel Syndrome
Keywords: mechanical interference; neural mobilization; ulnar neuropathy; post cubital syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome; Ulnar Neuropathies

STUDY DESIGN:
Intervention Model Description: mechanical interference and neural mobilization
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical interference (Experimental): the patients will receive mechanical interference and conventional treatment three times a week for four weeks
  Interventions: Other: Mechanical interference; Other: conventional treatment
- Neural mobilization (Experimental): the patients will receive neural mobilization and conventional treatment three times a week for four weeks
  Interventions: Other: Neural mobilization; Other: conventional treatment
- conventional treatment (Active Comparator): the patients will receive conventional treatment only three times a week for four weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Mechanical interference — The patients will receive mechanical interference treatment in the form of five techniques, including wrist distraction (3 sets for 3 minutes), rhythmic and gentle stretching of the transverse carpal ligaments, the release of palmar hand fascia, gliding of the finger flexor tendons (using the oscillatory flexion-extension movement of the metacarpophalangeal joint) and release of the upper forearm muscle and fascia were applied. Manual techniques were performed total of 15 minutes in each session each technique included 3 sets for 3 minutes and conventional treatment
  Arms: Mechanical interference
Other: Neural mobilization — the patients will receive neurodynamic mobilizations, including sliding techniques and tensioning techniques which are thought to enhance ulnar nerve gliding and restore neural tissue mobility and conventional treatment
  Arms: Neural mobilization
Other: conventional treatment — the patients will receive therapeutic ultrasound (frequency of 1 MHz, intensity of 1 W/cm2, for 5 minutes), transcutaneous electrical nerve stimulation (TENS) (frequency of 80 Hz, pulse duration of 60 μs, at the level of comfortable tingling sensation, for 20 minutes) and therapeutic exercises.

SUMMARY:
this study will be conducted to compare between mechanical interference and neural mobilization on ulnar neuropathy post-cubital tunnel syndrome

DETAILED DESCRIPTION:
Ulnar nerve neuropathies are the second most common entrapment neuropathy of the upper extremities after carpal tunnel syndrome. Cubital tunnel syndrome (CTS) is a condition that involves pressure or stretching of the ulnar nerve also known as the "funny bone" nerve, which could cause numbness or tingling in the ring and tiny fingers, pain in the forearm, and hand weakness. The ulnar nerve runs in a groove on the inner side of the elbow. Conservative treatment of cubital tunnel syndrome is recommended for patients with mild and moderate symptoms and without changes in cutaneous sensation or muscle atrophy. In addition, a wide variety of conservative approaches including corticosteroid injections as a minimally invasive technique and splinting and bracing failure were recommended for CTS depending on its severity. Manual therapy techniques are part of the physical therapy treatment of CTS, which are classified into two groups including nerve mobilization and mechanical interface mobilization. The aim of the study was to find which manual therapy method-technique directed to mechanical interface and nerve mobilization-has superior beneficial effects on clinical and electrophysiological findings in the conservative management of patients with CTS. Ninety patients with post-cubital syndrome will be allocated randomly to three groups; the first experimental one will receive mechanical interference, the second experimental will receive neural mobilization and the third one will receive conventional treatment for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed and referred by an orthopedist.
* The patient's age ranged from 20 to 55 years old.
* Recent NCV for ulnar nerve confirming the diagnosis.
* Unilateral cubital tunnel syndrome with ulnar neuropathy

Exclusion Criteria:

* Patients with cervical brachialgia.
* Patients with metabolic diseases such as diabetes, severe thyroid disorders, anemia, and -pregnancy.
* Hypertensive patients or patients who had a previous hand or elbow surgery.
* Patients with median nerve involvement in proximal areas such as thoracic outlet syndrome.

History of carpal tunnel release surgery. Steroid injection

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  pain will be measured by visual analogue scale. it is a vertical or horizontal 100mm line graduated by different level of pain, starting from 0 (no pain) till 100 (worst pain).

SECONDARY OUTCOMES:
function and severity | up to four weeks
  Boston Questionnaire will be used for assessing the function and severity of hand. The questionnaire including two parts, namely the symptom severity scale (SSS) and the functional status scale (FSS), is considered a standard tool to evaluate the patients with CTS. The SSS contains 11 questions on different symptoms of hand and FSS comprises of 5 questions assessing the difficulty in performing selected activities. The response to each question was scored from one (mildest) to five (most severe) points. The overall scores for SSS and FSS were calculated as the score sum of all questions.
ulnar nerve sensory conduction velocity | up to four weeks
  electromyography device will be used for measuring ulnar nerve sensory conduction velocity
ulnar nerve motor distal latency | up to four weeks
  electromyography device will be used for measuring ulnar nerve motor distal latency